CLINICAL TRIAL: NCT05531513
Title: The Effects of a Nature-Based Mindfulness-Compassion Intervention for Older Adults Delivered Using Virtual Reality: A Randomized Controlled Trial
Brief Title: The Effects of a Nature-Based Mindfulness-Compassion Intervention for Older Adults Delivered Using Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Super Sublime | Super Splendide (Unknown); Résidences Enharmonie (Unknown)
Responsible Party: Principal Investigator, Bassam Khoury, PhD, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: McGill University
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Mental Health Wellness 1; Healthy Aging
Keywords: virtual reality; nature; mindfulness; compassion; Gerontechnology; well-being; mental health; older adults
MeSH Terms: conditions — Psychological Well-Being | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: After providing consent, potential participants will complete an initial screening with the demographic intake form. Participants who do not meet inclusion or exclusion criteria will be informed that they will be unable to participate in the current study. Participants who meet study criteria will then be asked to complete the baseline survey containing the battery of outcome measures. Upon completion of the baseline measures, participants will be randomly assigned to one of two conditions: the experimental (Virtual Reality) condition or the active control (Psychoeducational Pamphlet) condition. Randomization will occur using a computerized random number generator following a matched random assignment via block procedure. An individual at arm's length (not involved with the intervention, assessment, or analysis) will perform the randomization. Control group participants will be allowed access to the virtual reality program after follow-up data collection is completed (after Week 9).
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to baseline assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (VR) Meditation (Experimental): The VR Meditation intervention will be administered in Arm 1.
  Interventions: Behavioral: Virtual Reality (VR) Meditation
- Psychoeducational Pamphlets (Active Comparator): The Psychoeducation Pamphlet intervention will be administered in Arm 2.
  Interventions: Behavioral: Psychoeducational Pamphlet

INTERVENTIONS:
Behavioral: Virtual Reality (VR) Meditation — The VR-Meditation intervention comprises an evidence-based 360-degree high-definition video VR application incorporating elements of nature, mindfulness and compassion. The VR-Meditation intervention is 4 weeks long and includes includes 4 different themes during the course of the program. Each week will focus on a distinct theme and will consist of two 20-minute VR sessions starting with a 10-minute guided meditation related to the weekly theme (one new meditation per week), followed by 10 minutes of open exploration of the virtual environment, for a total of 8 distinct sessions. The weekly themes are as follows:
  * Week 1 - Mindfulness of the Environment
  * Week 2 - Embodied Mindfulness
  * Week 3 - Embodied and Embedded Compassion
  * Week 4 - Mindfulness, Compassion, and the External Environment
  In addition to baseline measures, participants in the VR Meditation condition will be asked to complete measures at mid-point (week 3), post-intervention (week 5), and follow-up (week 9).
  Other Names: Toujours Dimanche
  Arms: Virtual Reality (VR) Meditation
Behavioral: Psychoeducational Pamphlet — The Psychoeducational Pamphlet intervention is 4 weeks long. Participants receive 1 pamphlet per week for a total of 4 different pamphlets. Handouts will provide information about managing stress and enhancing well-being, without referencing nature, mindfulness or compassion (e.g., eating habits, sleep hygiene, relaxation training, art exercises). The handouts will be based on empirical findings and will be written in accessible language with visual charts and specific practices to facilitate their implementation by participants. At the end of the study (i.e., after follow-up), Psychoeducation Pamphlet participants will receive access to the VR-Meditation program.
  In addition to baseline measures, participants in the Psycho-educational Pamphlet condition will be asked to complete measures at mid-point (week 3), post-intervention (week 5), and follow-up (week 9).
  Arms: Psychoeducational Pamphlets

SUMMARY:
The global population is aging at an unprecedented rate, increasing the necessity for effective interventions targeting the mental health needs of older adults. Virtual reality (VR) is a type of technology with the potential to improve mental health and well-being that allows users, via electronic devices such as headsets or goggles, to interact within simulated environments. VR programs using nature, mindfulness-meditation, and compassion may be more immersive and engaging, with research showing that these programs are effective at improving mental health and well-being outcomes in younger adults. However, evidence in this area for older adults is currently lacking.

The present project intends to pilot and examine a multi-user 360-High Definition (HD) video VR application, called "Toujours Dimanche", developed in partnership with Super Sublime, a Montreal-based not-for-profit company. This VR application aims to support older adults through incorporating elements of nature, mindfulness-meditation, and compassion via a 4-week program of twice weekly, 10 to 20-minute meditation sessions, for a total of 8 sessions. Thus, this study seeks to pilot, revise and iteratively evaluate, via randomized control trial (RCT) methodology, the acceptability, feasibility, and effectiveness of a multi-user 360-HD video VR application (Toujours Dimanche) at improving older adult mental health and well-being.

It is hypothesized that engagement with the 4-week VR-Meditation intervention will lead to lower scores on stress and negative affect and improved scores on well-being, positive affect, and mindfulness, in addition to increased scores on coping self-efficacy, connection with nature, embodied mindfulness, and self-compassion, over time and as compared to the active control group (who will receive psycho-educational pamphlets 1x/week for 4 weeks).

DETAILED DESCRIPTION:
INTRODUCTION:

There is a need for effective health strategies to help older adults' psychological well-being; thus, the proposed study seeks to better understand how to support older adults' mental health through the use of a virtual reality (VR)-based nature, mindfulness-and-compassion meditation intervention.

Technology developed to meet older adults' quality of life needs, or Gerontechnology has been increasingly integrated into daily life routines and may have the potential to ameliorate treatment accessibility and quality. However, to maximize the effectiveness of these technology-based modalities, it is necessary to move beyond conventional telehealth methodologies and investigate fresh modalities of mental health provision for older adults, such as VR.

One way proposed to utilize VR 360-degree video technology most effectively is through the incorporation of natural settings in the VR experience. A growing body of research highlights the therapeutic efficacy of 360-degree nature videos, pointing to nature-based VR's capability to rapidly improve mood, as well as its potential to decrease physiological stress levels and enhance cognitive functioning.

Additionally, through its capacity to capture participants' attention and provide users the illusion of "being there" in the 3D computer-generated environment, VR may be particularly effective when incorporating mindfulness-based activities. Mindfulness can be described as the process of purposefully, and with acceptance, paying attention non-judgmentally to the present moment. By providing people with an interesting setting to practice mindfulness (e.g., simulated natural settings), limiting distractions from the real world, and increasing a sense of presence, VR may facilitate mindfulness practice. This is significant, given that mindfulness-based interventions (MBIs) are particularly suited to meet the needs of older adults. Together with mindfulness, self-compassion, defined as thinking, feeling, and acting kindly towards oneself, can be used as a complementary strategy in MBIs and has been shown to augment their effectiveness, with evidence linking self-compassion to improved well-being in later life.

Preliminary findings highlight that VR is a promising technology to support MBIs, with evidence pointing to an increase in well-being, self-compassion, and adherence among participants. However, to date, no study has tested mindfulness training using VR for older adults. Additionally, no study has looked at the combined effects of mindfulness training in natural settings using VR for older adults. The evaluation of a VR application with multi-user capability that incorporates evidence-based activities to improve well-being (e.g., nature, mindfulness, compassion) in older adults is thus a significant research-to-practice gap. Therefore, this study, with the support of an industry partnership with Super Sublime, aims to evaluate the feasibility and effectiveness of a multi-user VR-Meditation application (called Toujours Dimanche), at improving older adult well-being via nature-based mindfulness and compassion training. If this VR-Meditation program is found to be acceptable and satisfactory, as well as demonstrating actual effectiveness in enhancing older adult well-being, it will serve to promote positive mental health for older adults utilizing a technology that is accessible, and safe. The proposed project thus addresses a critical societal need by significantly enhancing older adults' capability to access natural settings, and engage in mindfulness and compassion techniques, through VR technology.

OBJECTIVES:

Compared to an active control group (Psychoeducational Pamphlet), to evaluate the feasibility and acceptability of a twice-weekly, 4-week VR-Meditation program, as well as its effects on stress, positive and negative affect, psychological well-being, mindfulness, coping self-efficacy, connection with nature, and self-compassion.

HYPOTHESIS:

It is hypothesized that engagement with the 4-week VR-Meditation intervention will lead to lower scores on stress and negative affect and improved scores on well-being, positive affect, and mindfulness, in addition to increased scores on coping self-efficacy, connection with nature, embodied mindfulness, and self-compassion, over time and as compared to the active control group (who will receive psycho-educational pamphlets 1x/week for 4 weeks).

METHODS:

In this RCT, we aim to recruit 30 participants aged 60 and over residing in private residences for autonomous older adults in the Montreal, Quebec area (under the administration of Résidences Enharmonie). Based on conventions set by Julious (2005) for pilot studies, 12 participants per group is the recommended sample size to assess intervention feasibility and refine estimates for use in larger scale efficacy trials. For the present study, 24 participants would need to be recruited to meet this recommendation. In order to account for attrition, we aim to recruit 30 participants, with support from the Résidences ENHARMONIE's team of recreation therapists.

Upon completion of the baseline measures, participants will be randomly assigned to one of two conditions: the experimental condition (VR-Meditation) or the active control condition (Psychoeducational Pamphlet).

Participants in the VR-Meditation condition will be asked to use the VR program for a period of 4 weeks (2 seated VR meditation sessions per week, approximately 20 minutes per session, total of 8 sessions). Participants will use Oculus Quest 2 VR Headsets for the meditation sessions and research assistants will guide participants' usage of the VR-Meditation app via Samsung Galaxy Tab S6 tablets.

Participants in the Psychoeducational Pamphlet group will receive weekly pamphlets for a total of 4 distinct pamphlets. Handouts will provide information about managing stress and enhancing well-being, without referencing nature, mindfulness or compassion (e.g., eating habits, sleep hygiene, relaxation training, art exercises). The handouts will be based on empirical findings and will be written in accessible language with visual charts and specific practices to facilitate their implementation by participants. Additionally, at the end of the study (i.e., after follow-up), Psychoeducation Pamphlet participants will receive access to the VR-Meditation program.

Both conditions will be asked to complete questionnaires at baseline (pre-participation; week 1), mid-point (week 3), post participation (week 5) and follow-up (week 9).

RESEARCH SETTING:

The experiment will take place in 2-3 private independent seniors' residences in the Montreal, Quebec area, managed by Residences Enharmonie, and in the presence of a trained co-researcher. The data collections will be conducted with the help of a trained co-researcher. The research team will also train the residence staff regarding how to use and monitor the VR headsets and to implement the Toujours Dimanche program with participants.

PROPOSED ANALYSIS:

Qualitative data will be analyzed using a process of recursive abstraction in order to summarize the information by theme. Descriptive statistics for continuous variables will include means and standard deviations, and categorical variables will be summarized using frequencies and proportions. Outcome measure scores will be compared between the intervention and control groups using a 2 x 4 mixed MANOVA with within-subject (time) and between-subject (group) factors. Correlational analyses will be used to assess the relationship between outcome variables at baseline. Additionally, multivariate analyses of covariance (MANCOVA) will be run controlling for baseline levels of mindfulness =and nature connectedness.

ELIGIBILITY:
Inclusion Criteria:

* Must reside at a Résidence Enharmonie private residence for autonomous older adults in the Montreal, Quebec region
* Must be 60 years of age or older
* Ability to speak English or French

Exclusion Criteria:

* History of recurrent migraines/seizures/Traumatic Brain Injury during the past year
* Glaucoma or recovery phase of any eye surgery
* Diagnosed epilepsy or severe vertigo

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Scores on the Perceived Stress Scale (PSS) | At baseline (week 1), mid-point (week 3), post-intervention (week 5) and follow-up (week 9)
  PSS is a 14-item scale used to measure the degree to which life events are experienced and appraised as stressful. It asks respondents how often they have felt certain ways in the past month, with responses ranging from 0 (never) to 4 (very often). English and French versions available.
Change from Baseline in Scores on the Scale of Positive and Negative Experience (SPANE) | At baseline (week 1), mid-point (week 3), post-intervention (week 5) and follow-up (week 9)
  SPANE is a 12-item questionnaire with six items to assess positive feelings and six items to assess negative feelings. Participants are asked to rate their levels of affect using a 5-point scale ranging from 1 (rarely or never) to 5 (very often or always). English and French versions available.
Change from Baseline in Scores on the Flourishing Scale (FS) | At baseline (week 1), mid-point (week 3), post-intervention (week 5) and follow-up (week 9)
  The FS is a brief 8-item measure assessing participants' self-perceived success (e.g., purpose, self-esteem, relationships, optimism) and provides a single psychological well-being score. Participants are asked to rate their levels of well-being on a 7-point scale ranging from 1 (strongly disagree) to 7 (strongly agree). English and French versions available.
Change from Baseline in Scores on the General Self-Efficacy Scale (GSE) | At baseline (week 1), mid-point (week 3), post-intervention (week 5) and follow-up (week 9)
  The GSE is a 10-item scale that measures an individual's confidence in their ability to effectively cope with life challenges. Participants are asked to rate statements on a 4-point scale ranging from 1 (not at all true) to 4 (exactly true). English and French versions available.

SECONDARY OUTCOMES:
Change from Baseline in Scores on the Five Facet Mindfulness Questionnaire-Short Form (FFMQ-24) | At baseline (week 1), mid-point (week 3), post-intervention (week 5) and follow-up (week 9)
  The FFMQ-24 is a 24-item self-report measure derived from the longer 39-item measure assessing five specific facets of mindfulness: acting with awareness, describing, observing, non-reactivity, and non-judgmental acceptance. Participants rate their responses on a 5-point scale ranging from 1 (never or very rarely true) to 5 (very often or always true). English and French versions available.
Change from Baseline in Scores on the Connectedness to Nature Scale (CNS) | At baseline (week 1), mid-point (week 3), post-intervention (week 5) and follow-up (week 9)
  The CNS is a 14-item measure assessing individuals' sense of "oneness" with their natural environment. Items are rated on a 5-point scale ranging from 1 (strongly disagree) to 5 (strongly agree). English and French versions available.
Change from Baseline in Scores on the Embodied Mindfulness Questionnaire (EMQ) | At baseline (week 1), mid-point (week 3), post-intervention (week 5) and follow-up (week 9)
  The EMQ is a 24-item questionnaire assessing five dimensions of individual levels of embodied mindfulness: detachment from automatic thinking, awareness of the body, connection with the body, awareness of the mind-body connection, and acceptance of feelings and bodily sensations. Participants rate their responses on a 5-point scale ranging from 1 (almost never) to 6 (almost always). English version only.
Change from Baseline in Scores on the Self-Compassion Questionnaire-Self (CQS) | At baseline (week 1), mid-point (week 3), post-intervention (week 5) and follow-up (week 9)
  The CQS is a newly developed 20-item questionnaire that assesses individual levels of self-compassion and is based on thinking, feeling, acting, and interpersonal components. Participants rate their responses on a 5-point scale ranging from 1 (almost never) to 5 (almost always). English version only.

OTHER OUTCOMES:
Change from Time 1 in Scores on the Simulator Sickness Questionnaire (SSQ) | After the first VR Meditation session at time 1 (week 2), mid-point (week 3), and post-intervention (week 5)
  The SSQ is a 16-item scale that is widely used to assess simulator sickness. The SSQ will only be administered to participants in the VR Meditation condition.
Researcher Developed Virtual Reality Program Satisfaction Questionnaire | Post-intervention (week 5)
  Participants in the VR Meditation condition will be asked a series of structured and open-ended questions at the end of their final VR session (session 8, week 5). The structured questions will involve a rating scale of 1-6 ranging from 1 (strongly disagree) to 6 (strongly agree). Questions will examine participant success in navigating the program, their enjoyment, their discomfort, and whether they would be likely to use the program again, as well as whether they perceived any changes in their meditation practices, relationship with nature, and relationship with technology.

CONTACTS AND LOCATIONS:
Overall Officials: Bassam Khoury, PhD, Principal Investigator — McGill University
Locations (2):
- Canada (2):
  - Piero Corti Residence, Montreal, Quebec
  - Résidences Enharmonie - Résidence Alfredo-Gagliardi, Montreal, Quebec